CLINICAL TRIAL: NCT01223430
Title: Simultaneously Using Traditional Chinese Medicine (Si-Ni-Tang) to Treat Septic Shock Patients - a Double Blind, Prospective, Randomized Controlled Study
Brief Title: Simultaneously Using Traditional Chinese Medicine (Si-Ni-Tang) to Treat Septic Shock Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The IRB considered our trial risky. Although there were debates between investigators and IRB, we terminated our trial in accordance with the suggestion of IRB.
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Huang-Chi Chen, Attending Physician of the Internal Medicine Department, Changhua Christian Hospital, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCH IRB 100105
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Septic Shock
Keywords: septic shock; shock reversal; ICU; traditional Chinese medicine
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Si-Ni-Tang (Experimental)
  Interventions: Drug: Si-Ni-Tang/ Placebo of Si-Ni-Tang
- Placebo (Placebo Comparator)
  Interventions: Drug: Si-Ni-Tang/ Placebo of Si-Ni-Tang

INTERVENTIONS:
Drug: Si-Ni-Tang/ Placebo of Si-Ni-Tang — The prescription is 2.25 grams four times a day ( 9 grams per day) for 7 days or till shock reversal( if shock reversal < 1 week). Shock reversal was defined as the discontinuation of norepinephrine or dopamine lasting for at least 24 hours.

SUMMARY:
The purpose of this study is to determine whether simultaneously using the traditional Chinese medicine, Si-Ni-Tang, is more effective in the treatment of septic shock patients.

DETAILED DESCRIPTION:
Those with hemodynamic instability were the main population of the ICU patients, whether the exact etiology leading to the diseases. However, how to maintain adequate hemodynamic status in order to keep the patients with well organs perfusion is the main issue of the intensive care physicians. The choices of vasoactive drugs in the guidelines or experts' suggestions nowadays used are still limited in the western medicine. Si-Ni-Tang, a remedy previously used in ancient China and now widely prescribed in Taiwan and China, is used for treating patients diagnosed as shock or heart failure. The investigators are eager to know if there existed any benefit via adding this drug to treat the septic shock patients. Therefore, the investigators designed a prospectively randomized double blind control trial to determine whether simultaneously using the traditional Chinese medicine, Si-Ni-Tang, is more effective in the treatment of septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to our intensive care units are enrolled if their disease diagnosis meets the definition of septic shock
* Using vasopressor now and the duration from initiation of vasopressor use to the entrance of the study is within 24 hours
* Nasogastric tube feeding

Exclusion Criteria:

* More than one kind of vasopressor is administrated
* Patients with extremely poor gastrointestinal function and can not tolerate diet feeding
* Acute myocardial infarction
* Patients with evidence of major bleeding
* Expected surgical intervention or scheduled surgery in the subsequent one week
* Patients who received digoxin for arrhythmia in the past one week

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
time to cessation of vasopressor use | one week

SECONDARY OUTCOMES:
intensive care unit (ICU) mortality | one month
ICU length of stay | one month
28-day survival rate | one month

CONTACTS AND LOCATIONS:
Overall Officials: Huang-Chi CHEN, M.D., Principal Investigator — Changhua Christian Hospital, TAIWAN
Locations (1):
- Medical ICU, Changhua Christian Hospital, Changhua, Taiwan, Taiwan

REFERENCES:
- [Derived] Chen HC, Chen WC, Lin KH, Chen YH, Lo LC, Lee TC, Hsia TC, Wang CH, Wu SH, Hsu HW, Chang YJ, Huang YC, Ku TH, Horng MH. Simultaneous use of traditional Chinese medicine (si-ni-tang) to treat septic shock patients: study protocol for a randomized controlled trial. Trials. 2011 Aug 24;12:199. doi: 10.1186/1745-6215-12-199. PMID 21864392